CLINICAL TRIAL: NCT01392235
Title: A Single-arm, Open, Multicenter, Phase II Study of Famitinib as ≥Third Line Treatment in Patients With Recurrent and/or Metastatic Nasopharyngeal Carcinoma (NPC)
Brief Title: Famitinib in Treating Patients With Recurrent and/or Metastatic Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTN-II-NPC
Record Dates: First submitted 2011-07-03; First posted 2011-07-12 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2018-12

CONDITIONS: Recurrent Nasopharyngeal Carcinoma; Metastatic Nasopharyngeal Carcinoma
Keywords: Recurrent and/or Metastatic Nasopharyngeal Carcinoma (NPC)
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug: Famitinib (Experimental)
  Interventions: Drug: Famitinib

INTERVENTIONS:
Drug: Famitinib — 25 mg qd p.o. and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
RATIONALE: Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3. Phase I study has shown that the drug's toxicity is manageable.

PURPOSE: This phase II trial is studying how well famitinib works in treating patients with recurrent and/or metastatic NPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologic confirmed recurrent and/or metastatic nasopharyngeal carcinoma( NPC )
* Have failed for ≥2 lines of chemotherapy
* At least one measurable lesion, larger than 10 mm in diameter by spiral CT scan(scanning layer ≤ 5 mm )
* ≥ 18 and ≤ 70 years of age
* ECOG performance scale 0-2
* Life expectancy of more than 3 months
* More than 4 weeks after operation, chemotherapy, radiotherapy, cytotoxic agents or tyrosine kinase inhibitors
* Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥ 90g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, 24-hour urinary protein ≤ 1.0 g total bilirubin < 1.25×the upper limit of normal(ULN), and serum transaminase < 1.5×the ULN (If liver metastases, serum transaminase< 2.5×the ULN), serum creatine ≤ 1x ULN, creatinine clearance rate > 50ml/min, Cholesterol≤7.75 mmol/L and triglyceride≤2.5 x ULN, LVEF: ≥ 50%
* Patients could provide 4-6 pieces of organization wax or pathological section
* Female: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article. Child bearing potential, a negative urine or serum pregnancy test result before initiating Famitinib. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article.
* Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Prior therapy with tyrosine kinase -inhibitor agent targeting at VEGFR, PDGFR and c-Kit
* Prior radiotherapy more than 2 courses
* Before or at the same time any, second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Less than 4 weeks from the last clinical trial
* Any factors that influence the usage of oral administration
* Known Spinal Cord compression or diseases of brain or pia mater by CT /MRI screening
* Imageology shows that tumor lesion less than 5 mm to great vessels
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg despite using single medical therapy, more than cla ss I (NCI CTCAE 3.0 ) myocardial ischemia, arrhythmia, or cardiac insufficiency
* URT: urine protein ≥ ++ and > 1.0 g of 24 h
* Long-term untreated wounds or fractures
* Blood coagulation abnormal, having hemorrhagic tendency (eg. active peptic ulcer disease) or receiving the therapy of thrombolysis or anticoagulation.
* Within 6 months before the first treatment occurrs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc.
* Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; If the prothrombin time international normalized ratio (INR) ≤ 1.5, with the purpose of prevention, the use of small doses of warfarin (1mg orally, once daily) or low-dose aspirin (between 80mg to 100mg daily) is allowed
* Preexisting thyroid dysfunction, even using medical therapy, thyroid function cannot maintain in the normal range
* Abuse of Psychiatric drugs or dysphrenia
* Viral hepatitis type B or type C
* Immunodeficiency: HIV positive, or other acquired immunodeficiency, congenital immunodeficiency, or organ transplantation
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
CBR(Clinical Benefit Rate) | 12 weeks
  To evaluate the efficacy (clinical benefit rate) of single-agent famitinib in patients with recurrent or metastatic NPC

SECONDARY OUTCOMES:
ORR (Objective Response Rate) | 12 weeks
PFS(Progress Free Survival) | 3 years
DCR(Disease Control Rate) | 12 weeks
OS(Sverall Survival) | 3 years
To evaluate the safety and tolerability | 3 years
  Number of participants with adverse events and serious adverse events.In addition,estimating their relationship with Famitinib.
QoL(Quality of Life) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Cancer Center, Sun Yet-sen University, Guangzhou, Guangdong, China